CLINICAL TRIAL: NCT02026362
Title: Randomized, Open-label, Multi-center Clinical Trial to Compare the Efficacy and Safety of MASCT Group' and 'Non-treatment Group' in Patient Undergone Curative Resection( RFA or Operation) for Hepatocellular Carcinoma .MASCT That Expresses Multiple Antigens Specific Cellular Therapy,Autologous Immune Cytotoxic of T-lymphocytes(CTL) Induced by Dendritic Cell(DC) Loaded With Multiple Antigens
Brief Title: Multiple Antigen Specific Cell Therapy (MASCT) for Hepatocellular Carcinoma(HCC) Patients After Radical Resection or Radio Frequency Ablation(RFA).
Acronym: HCC DC CTL
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Interim analysis
Sponsor: HRYZ Biotech Co. (Industry)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-sen University (Other); Beijing 302 Hospital (Other); Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYZ Cell Therapy Co..
Record Dates: First submitted 2013-12-11; First posted 2014-01-03 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; DC; CTL
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The foundation treatment after radical operation or RFA (Other): The foundation treatment including against hepatitis b virus treatment using nucleoside analogue drug and protect liver treatment
  Interventions: Other: The foundation treatment including against hepatitis b virus treatment using nucleoside analogue drug and protect liver treatment
- MASCT:Multiple Antigens Specific Cellular Therapy (Experimental): autologous immune cytotoxic of T-lymphocytes (CTL) induced by dendritic cells, (DC) loaded with multiple antigens DC loaded with survivin p53 her2 ect total 17 antigens
  Interventions: Biological: MASCT:Multiple Antigens Specific Cellular Therapy; Other: The foundation treatment including against hepatitis b virus treatment using nucleoside analogue drug and protect liver treatment

INTERVENTIONS:
Biological: MASCT:Multiple Antigens Specific Cellular Therapy — autologous immune cytotoxic of T-lymphocytes (CTL) induced by dendritic cells, (DC) loaded with multiple antigens DC loaded with survivin p53 her2 ect total 17 antigens .
  Arms: MASCT:Multiple Antigens Specific Cellular Therapy
Other: The foundation treatment including against hepatitis b virus treatment using nucleoside analogue drug and protect liver treatment

SUMMARY:
To prove that the efficacy and safety of 'MASCT group' is superior to 'non-treatment group' in patient undergone curative resection (RFA or operation) for hepatocellular carcinoma in China.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is diagnosed as hepatocellular carcinoma(HCC);
2. The patient underwent radical operation of HCC within 8 weeks before enrollment;
3. The number of tumors≤2；
4. No cancer embolus in the main portal vein and first branch, hepatic duct and first branch, hepatic vein, inferior vena cava;
5. No portal lymph node metastasis；
6. No extra-hepatic metastasis;
7. Complete tumor resection without residual tumor at the surgical margins should be confirmed by enhanced CT or MRI imaging within 4 week (including 4 weeks) after radical operation;
8. If an increased serum AFP level was detected of the patient before the radical operation, the AFP level should be returned to normal in 8 weeks;
9. Child-Pugh Score ≤9;
10. ECOG Performance status (ECOG-PS) ≤2 ;
11. The expected survival time > 2 years;
12. Tests of blood,liver and kidney should meet the following criteria：

    * WBC>3×109/L
    * Neutrophil counts >1.5×109/L
    * Hemoglobin ≥85 g/L
    * Platelet counts≥50×109/L
    * PT is normal or The extend time <3s
    * BUN≤1.5 times the upper-limit ,
    * Serum creatinine≤ 1.5 times of the upper-limit
13. Sign the informed consent.

Exclusion Criteria:

1. Women who is pregnant or during breast feeding or plan to pregnant in 2 years;
2. Extra-hepatic metastasis or liver residual tumor;
3. Cancer embolus in the main portal vein and first branch, Hepatic duct and first branch, hepatic vein, inferior vena cava;
4. 6 months before enrollment: the period of systemic and continuous use of immunomodulatory agents (such as interferon, thymosin, traditional Chinese medicine) was longer than 3 months;
5. 6 months before enrollment: the period of systemic and continuous use of the immunosuppressive drugs (such as corticosteroids drug) was longer than 1 months;
6. Received any cell therapy (including NK, CIK, DC, CTL, stem cells therapy) in 6 months before enrollment;
7. Positive for HIV antibody or HCV antibody;
8. Have a history of immunodeficiency disease or autoimmune diseases (such as rheumatoid arthritis, Buerger's disease, multiple sclerosis and diabetes type 1);
9. Patient who suffered from other malignant tumor in 5 years before enrollment (except skin cancer, localized prostate cancer or cervix carcinoma);
10. . Patients with organ failure;
11. Patients with serious mental disease;
12. Drug addiction in 1year before enrollment (including alcoholics);
13. Participated in other clinical trials in 3 months before screening;
14. Other reasons the researchers think not suitable.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-07 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with tumor recurrence or metastasis | 5years
Time of tumor recurrence or metastasis | 5 years

SECONDARY OUTCOMES:
Hepatitis B virus markers figures | an expected average of 18 weeks
Serum hepatitis B virus (HBV)DNA figures | an expected average of 16 weeks
overall survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- JOE ZHOU, Shenzhen, Guangdong, China

REFERENCES:
- See also: Related Info — http://www.nfyy.com/
- See also: Related Info — http://www.sysucc.org.cn/
- See also: Related Info — http://www.zssy.com.cn/